CLINICAL TRIAL: NCT03650907
Title: Exercise Intervention for Patients With Sarcopenia or Frailty in Long-term Care Institutions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wen-Chun Tseng, Physiatrist, Physical Medicine and Rehabilitation, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SarcExercise
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group exercise program by coach (Experimental)
  Interventions: Behavioral: Group exercise program
- Self exercise (Sham Comparator)
  Interventions: Behavioral: Self exercise program

INTERVENTIONS:
Behavioral: Group exercise program — Patients in experimental group attend group exercise program, instructed by fitness trainer, at long-term care institutions.
  Frequency: 3 times per week. Type: resistance/flexibility/balance training, including warm-up and cold-down. Duration: 1 hour per time, for 16 weeks.
  Arms: Group exercise program by coach
Behavioral: Self exercise program — Patients in control group receive oral education for self exercise program, mainly resistance muscle training. Patients are requested to do self-training for 16 weeks.
  Arms: Self exercise

SUMMARY:
Sarcopenia is a geriatric syndrome of decreased muscle volume with muscular function decline. There is more tendency for sarcopenic elderly to be frail, disabled, or have cardiovascular disease. Compared to those who are not sarcopenic, they also had worse prognosis in response to treatment for definite diseases, and spend more medical cost.

Exercise appears to have an important role in management of sarcopenia. In the current study, the investigators provide an exercise program, including resistance/balance training for the elderly with sarcopenia or frailty in long-term care institution, and evaluate the effect.

ELIGIBILITY:
Inclusion Criteria:

1. >20-year-old
2. diagnosed with sarcopenia (by the definition from Asia workgroup for sarcopenia, AWGS) or frailty (The Fried model, based on five functional criteria)

Exclusion Criteria:

1. Severe medical diseases or mental problems, which result in difficulty to follow exercise program.
2. Inability to get down from bed for activity due to disease, such as neuropathy or orthopedic disease.
3. High risk group for exercise program, such as those with unstable fracture or nonunion fracture.
4. Anyone who didn't want attend this study.

Ages: 20 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Muscle strength | after 16-weeks training
  grasp strength by dynamometer
walk speed | after 16-weeks training
  6-meter walk test

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chun Tseng, Principal Investigator — Chang Gung Medical Hospital
Locations (1):
- Bor-Ay Sweet home, Keelung, Taiwan